CLINICAL TRIAL: NCT01116063
Title: Inhaled Iloprost for Disproportionate Pulmonary Hypertension in Chronic Obstructive Pulmonary Disease
Brief Title: Inhaled Iloprost for Disproportionate Pulmonary Hypertension in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPDVEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Yochai Adir, Director pulmonary hypertesnion service, Pulmonary divison Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COPDVEN 2009
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Pulmonary hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm open label (Experimental): All patients will receive the study drugs and will be evaluated
  Interventions: Drug: Inhaled iloprost

INTERVENTIONS:
Drug: Inhaled iloprost — Inhalation Initial: 2.5 mcg/dose; if tolerated, increase to 5 mcg/dose; administer 6 times daily
  Other Names: Brand name - Ventavis

SUMMARY:
Pulmonary hypertension is frequently present in COPD and it is generally limited to a mild increase in mean pulmonary artery pressure. However some COPD patients are characterized by higher levels of mPAP at rest, fulfilling the definition of moderate or severe PH disproportionate PH .

In these patients the elevated pulmonary pressures adversely affect the prognosis.At the present time the evidence for the the use of specific pulmonary vasodilators in the management of these patients are scarce and cannot be recommended.the aim of this study is to evaluate the medium term efficacy and safety of the inhaled prostacyclin stable analog, iloprost in patients with COPD and moderate to severe pulmonary hypertension

DETAILED DESCRIPTION:
While pulmonary hypertension is frequently present in COPD, particularly in the presence of hypoxemia, it is generally limited to a mild increase in mean pulmonary artery pressure in the face of a normal cardiac output.

Apart from this classical and widely observed profile of PH with modestly elevated mPAP, some COPD patients are characterized by higher levels of mPAP at rest, fulfilling the definition of moderate or severe PH . This kind of PH may be observed in patients presenting with a severe obstructive disease, but sometimes contrasts with a mild or moderate obstruction. In the latter case, the term disproportionate PH has been proposed, but it can be extended to describe all COPD patients with moderate to- severe PH.

Therefore, it is possible that in some patients with COPD, pulmonary hypertension contributes to the clinical picture because of right ventricular output limitation and is responsible for the poor prognosis of these patients, which is similar to that in primary pulmonary arterial hypertension.

The exact incidence of clinically significant pulmonary hypertension, defined as pulmonary hypertension that contributes to symptomatology and prognosis, is difficult to estimate in COPD. A prevalence of 5.8%- 13.5% in patients seems reasonable which would suggest an incidence of 1-3/10,000, which is 100 times the incidence of idiopathic pulmonary arterial hypertension.

These patients are characterized by marked effort dyspnea , profound hypoxemia, hypocapnia, moderate airway obstruction and a very low DLCO.

PH in COPD was an independent prognostic factor. Indeed, patients with similar airflow limitation had lower life expectancy when PH was resent. Patients with PH had a significantly lower survival rate at 5 yrs compared with patients without PH (33 versus 66%). Pathologic studies that stemmed from long-term oxygen trials pointed to the fact that pulmonary vascular remodeling in chronic obstructive pulmonary disease (COPD) is more than just medial hypertrophy from long-lasting hypoxic vasoconstriction. In these patients, all vessel wall layers appear to be involved, with intimal changes actually being the most prominent. Major remodeling of all pulmonary arterial vessel layers explains why pulmonary hypertension in COPD is often not,or minimally, reversible by supplemental oxygen, acutely or chronically. The pathobiology of pulmonary artery remodeling in advanced COPD remains incompletely explored. There are data supporting an endothelium-derived vasoconstrictor-dilator imbalance, mainly from a decreased endothelial nitric oxide expression. Plasma levels of ET-1 are increased both in patients with severe COPD and there is evidence that ETA and ETB receptor expression is increased in the pulmonary arteries of patients with COPD.

The major unmet medical need is the absence of a simple drug therapy that relieves the breathlessness or muscle fatigue, reduces pulmonary vascular resistance and the overloaded right ventricles that severely limits exercise tolerance in COPD and affects survival.

The only validated therapeutic approach of the 'common' PH in COPD patients is long-term oxygen therapy. A large variety of vasodilators has been tested in numerous studies both after short- and medium-term administration. The early enthusiasm vanished subsequently for several reasons: modesty of the vasodilator effect, inability for some drugs to sustain the acute benefit, no specificity of the vasodilator effect with concomitant systemic vasodilatation, deleterious effect on gas exchange due to a diminution of the ventilation/perfusion ratio and no demonstration of a survival benefit. At the present time vasodilators cannot be recommended in the management of COPD.

Treatments of PAH have shown a dramatic change in the past few years. Synthetic prostacyclin (epoprostenol), prostacyclin analogues, endothelin-1 receptor antagonists and phosphodiesterase-5 inhibitors are in use in group I PAH with improve clinical outcome.

Based on analogy to primary pulmonary hypertension, a specific interventions aiming at the restoration of endothelial vasoconstrictor- dilator imbalance could be undertaken.

Selective pulmonary vasodilatation by inhalation of the vasorelaxant agent is an appealing concept to circumvent some of the hazards inherent in systemic vasodilator therapy in COPD patients with PH. Treatment of these patients with aerosolization of iloprost may reduce pulmonary vascular resistance , increases cardiac output while conserving ventilation-perfusion matching and and shunt preventing worsening of arterial hypoxia and wasting of the small ventilatory reserve of these patients.

In order to resolve these uncertainties we suggest evaluating the effectiveness of an inhaled iloprost in COPD patients with moderate to severe pulmonary hypertension. This evaluation would include monitoring and measurement of all the relevant cardio-respiratory variables as set out in detail below.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with COPD and increased SPAP >55 on echocardiogram will be screened for the study.
2. Patients with normal wedge pressure ( [PCWP] ≤ 15 mm Hg), mean PAP ≥ 35 mm Hg and a pulmonary vascular resistance (PVR- 3.0 wood unit)on right heart catheterization.
3. Diagnosis of COPD according to GOLD guidelines
4. The patient can read, understand and sign the informed consent.

Exclusion Criteria:

1. Other identified cause for pulmonary hypertension

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance | 6 months

SECONDARY OUTCOMES:
6 minutes walking test | 6 months
Borg dyspnea score | 6 months
NT-BNP | 6 months
Arterial blood gases | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Adir, MD, Principal Investigator — Pulmoanry Division, Carmel Medical Center
Locations (1):
- Pulmoanry Division, Carmel Medical Center, Haifa, Israel